CLINICAL TRIAL: NCT04901143
Title: Meal Handling of Advanced Closed Loop Insulin Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Prof. Amir Tirosh, Prof. Amir Tirosh, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-21-8159-at-ctil
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Advanced hybrid closed loop system — Phase 1: meals in open loop- 3 weeks Phase 2: closed loop conventional meal announcement- 3 weeks Phase 3: closed loop, pre define universal bolus- 3 weeks

SUMMARY:
The study will Compare meal related glycemic indices following 2 types of meal announcement:

1. Conventional assessment of carb content plus carb equivalence of proteins and fat
2. Algorithm device optimal universal meal announce equivalent

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 20 to 70 years of age at time of screening
2. Subject's weight is between 50 and 120 kg
3. A clinical diagnosis of Type 1 diabetes as determined by the Investigator for a minimum of 36 months prior to enrollment
4. Subject has ongoing use of an insulin pump and rtCGM ≥ 6 months prior to screening
5. current use of 670G 4.0 pump
6. Subject has an A1C value ≤ 10.0% demonstrated at the time of enrollment.
7. Subject uses a rapid-acting analogue insulin in his/her pump
8. Patient is willing to undergo all study procedures
9. English proficiency
10. Minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units

Exclusion Criteria:

1. Female subject who has a positive serum pregnancy screening test, or who plans to become pregnant during the course of the study
2. Subject has unresolved adverse skin condition, or unable to tolerate tape adhesive, in the area of sensor placement or device replacement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject has a history of hypoglycemic seizure or hypoglycemic coma within the past 12 months
4. Subjects currently taking adjunct therapy with SGLT2-inhibitors, Amylin.
5. Subject has a history of seizure disorder unrelated to diabetes within the past 12 months
6. Gastroparesis, uncontrolled thyroid disorder, Addison disease,. , Pituitary insufficiency
7. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), congestive heart failure, ventricular rhythm disturbances, or thromboembolic disease within the past 6 months
8. Subject has a presence of a cardiac pacemaker or any other device that may be sensitive to radio frequency telemetry
9. Subject has any condition, including screening lab values that in the opinion of the Investigator may preclude him/her from participating in the study and completing study related procedures
10. Subject is actively participating in other investigational study (drug or device)
11. Subjects who consume alcohol daily
12. Use of CGM (other than per protocol) throughout the duration of the study
13. Use of Hydroxyurea medication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Time in range | 300 minutes
  AUC glucose 300 minutes post meal

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel